CLINICAL TRIAL: NCT03486561
Title: Management of Ischemic Heart Disease With Angiwell-XR (Ranolazine)
Acronym: MIDA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: OBS Pakistan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIDA-OBS-001
Record Dates: First submitted 2018-03-15; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Chronic Stable Angina
Keywords: Ranolazine; Pakistan; Ischemic Heart Disease
MeSH Terms: conditions — Angina, Stable; Myocardial Ischemia | interventions — Ranolazine

STUDY DESIGN:
Intervention Model Description: Open Labelled Phase IV clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ranolazine (Other): Ranolazine was approved by the U.S. Food and Drug Administration in 2006 in 500 mg and 1000 mg extended-release doses, advising 500 mg BID as a starting dose and 1000 mg BID as maximum dose
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine — Ranolazine inhibits sodium and potassium ion channel currents. Inhibition of the late phase of the inward sodium current during cardiac repolarization has been well studied4. In disease states, enhanced sodium-calcium exchange due to augmented late phase of the inward sodium current activity leads to increased cytosolic calcium concentration. Intracellular calcium overload is believed to be critical to the mechanism of decreased left ventricular relaxation caused by ischemia and reperfusion. Elevated left ventricular diastolic wall tension compromises myocardial blood flow even further.

SUMMARY:
The rationale of MIDA trial is to determine efficacy and tolerability of ranolazine molecule among Pakistan population and obtain firsthand knowledge about the molecule ranolazine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of coronary artery disease (CAD)

  * Patients present with the symptoms of stable angina after withdrawn from other antianginal drugs and given the required background therapy for at least 7 days will be qualified for entering this study and performing 1st ETT qualifying test
  * Patients developed exercise-induced ECG ischemiai during two qualifying exercise treadmill testsii.
  * Willing and able to provide a written informed consent

Exclusion Criteria:

* • Factors that might compromise ECG or ETT interpretation

  * Patients with resting ST-segment depression ≥ 1mm in any lead
  * Left bundle-branch block
  * Patients implanted with pacemaker
  * Patients under Digitalis therapy

    * Patients with family history of (or congenital) long QT syndrome
    * Patients with congenital heart disease
    * Patients with uncorrected valvular heart disease
    * Patients with unstable angina, or MI, or coronary revascularization procedure ≤ 2 months prior enter this study
    * Female who is pregnant/lactating or planning to be pregnant, or female of childbearing potential* who is not using medically recognized method of contraception
  * *Other than those who have been surgically sterilized (defined as having undergone hysterectomy or bilateral oophorectomy or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal.

    • Patients are under any one of the following conditions:
  * New York Heart Association (NYHA) Class III or Class IV congestive heart failure (CHF)
  * QTc > 450 msec at screening
  * Active myocarditis, pericarditis, hypertrophic cardiomyopathy
  * Uncontrolled hypertension (defined as SBP > 180 mmHg) Voltage criteria for left ventricular hypertrophy in the absence of repolarization abnormalities will not be exclusion criteria

    * Use of any investigational product ≤ 4 weeks prior to screening
    * Patients with severe hepatic disease (e.g., liver cirrhosis)
    * Patients with impaired renal function (defined as serum Cr >1.5 mg/dl)
    * Patients with any condition or disease which is considered not suitable for this study by investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Reduction in frequency of Angina with Ranolazine | 24 weeks
  To determine reduction in frequency of Angina with Ranolazine

SECONDARY OUTCOMES:
Safety: Proportion of participants experiencing an adverse event (AE) | 24 weeks
  Proportion of participants experiencing an adverse event (AE)

IPD SHARING:
Plan to Share IPD: No